CLINICAL TRIAL: NCT03697447
Title: Randomized, Controlled, Within-patient, Singleblind Study to Evaluate the Efficacy of 12-weeks of Endermotherapy With Adult Burn Survivors
Brief Title: Endermotherapy With Burn Hypertrophic Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15.374
Record Dates: First submitted 2018-03-22; First posted 2018-10-05 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Burn Scar

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endermotherapy treated scar (Experimental): Endermotherapy massage treatment
  Interventions: Procedure: Endermotherapy
- Control scar (No Intervention): No intervention, standard of care

INTERVENTIONS:
Procedure: Endermotherapy — Endermotherapy massage (mechanic massage) of burn scar
  Arms: Endermotherapy treated scar

SUMMARY:
Mechanical massage or endermotherapyTM is applied to scar tissue with the intended therapeutic value being the promotion of structural or physiological changes. These proposed changes are meant to induce more pliability, so that skin possesses the strength and elasticity required for normal mobility. The advantage of mechanical massage compared to manual massage is that it provides a standard dosage using rollers and suction valves to mobilize the tissue. However, research documenting and supporting this effect is lacking. The objective of this proposal is to document the effect of 12 weeks of endermotherapy treatment on hypertrophic scar characteristics, including erythema, pigmentation, pliability, and thickness in adult burn survivors and their subjective evaluation of itch, pain and overall scar outcome through a prospective, randomized, controlled, within-patient, single-blinded study.

DETAILED DESCRIPTION:
Patients will receive 12 weeks of endermotherapy , 3 times a week.

ELIGIBILITY:
Inclusion Criteria:

* females and males, of any race, 14 years or older,
* a thermal injury,
* at least 3 months post-burn so that the scars will be durable enough to tolerate the proposed forces,
* at least 2 scar sites >2.034 mm thick and within 0.5 mm of each other, and
* signed the informed patient consent form

Exclusion Criteria:

* subjects who have keloids,
* with a diagnosis of psychiatric illness clearly documented in their medical file,
* mechanism of injury is an electrical, chemical, or cold injury,
* a dermatological conditions in the region of the evaluation site, that may interfere with the study results,
* a suspected or known allergy to ultrasound gel,
* unable to understand French or English, or
* subjects who refuse to give informed consent.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Skin Thickness Changes | baseline, 12, 24 and 36 weeks
  Ultrasound skin measures, mm

SECONDARY OUTCOMES:
Cutometer Skin Elasticity Changes | baseline, 12, 24 and 36 weeks
  skin elasticity measures (r0- cutometer), mm
Mexameter Skin Erythema Changes | baseline, 12, 24 and 36 weeks
  Erythema index measure by Mexameter, scale values of 0 to 999. The erythema values are individual for each person and depend strongly on the ethnic group. The measurements are generally used to determine changes before and after a treatment.
Itch Visual Analog Subjective Changes | baseline, 12, 24 and 36 weeks
  Itch, Visual analog scale (score 0-none to 10-worse)
Pain Visual Analog Subjective Changes: VAS | baseline, 12, 24 and 36 weeks
  Pain, Visual analog scale (score 0-none to 10-worse)

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette Nedelec, PhD, Principal Investigator — CRCHUM
Locations (1):
- Montreal Burn Unit, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No